CLINICAL TRIAL: NCT02166099
Title: Choledochoscopy For Diagnosing Pancreatico-Biliary Disorders: A Multicenter Registry
Brief Title: Choledochoscopy Multicenter Registry
Acronym: SPY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief of Endoscopy, Weill Medical College of Cornell University
Other Study IDs: 1206012450
Record Dates: First submitted 2014-06-10; First posted 2014-06-18 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Pancreatico-biliary Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SpyGlass Choledochoscopy procedure: Any patient who has undergone SpyGlass Choledochoscopy procedures for diagnosis and/or treatment of a pancreatico-biliary disorder
  Interventions: Procedure: Choledochoscopy using Digital Spyglass

INTERVENTIONS:
Procedure: Choledochoscopy using Digital Spyglass — Choledochoscopy using Digital Spyglass during Endoscopy

SUMMARY:
The purpose of this registry is to record information and evaluate the impact of SpyGlassTM Direct Visualization System for choledochoscopy on the management of pancreatico-biliary disorders. The registry will evaluate diagnostic performance and overall clinical management impacted by SpyGlass.

This multi-center registry has been initiated:

* To document the impact of SpyGlass Choledochoscopy in pancreatico-biliary disorders on the clinical management of pancreatico-biliary disorders including malignancies.
* To assess the sensitivity, specificity, accuracy, technical feasibility, safety and cost effectiveness of SpyGlass and compare it to other diagnostic modalities.

DETAILED DESCRIPTION:
Our institution performs therapeutic Interventional Endoscopy in around 750-1000 patients a year. During these interventional procedures, advanced and emerging imaging techniques including choledochoscopy, choledochopancreatoscopy, confocal endomicroscopy, chromoendoscopy, narrow band imaging, etc. are conducted for presumptive or definitive diagnoses in some of the patients suffering pancreatico-biliary disorders; including malignancies. Early and accurate diagnosis is necessary to improve the prognosis for pancreatic cancer or cholangiocarcinoma. Initial studies have shown that advanced imaging including confocal microendoscopy may majorly impact the clinical management of patients by providing accurate diagnosis early on. Choledochoscopy is used for microendoscopic visualisation of lumen and mucous membrane, for diagnosis, classification and therapy of abnormally functioning gall-bladder and pancreatic systems. New refinements have allowed for single user direct imaging with endobiliary biopsy. SpyGlassTM Direct Visualization System (Boston Scientific, Natick, MA) is a platform designed to enhance diagnostic accuracy during ERCP (Endoscopic Retrograde Cholangiopancreatography) and allowing guided biopsy. It is an FDA approved instrument with the ability of performing cholangiopancreatoscopy by a single endoscopist during ERCP. A 1.2 mm working channel exists within the Spyglass system allowing for instrument access to the biliary or pancreatic tree. Advanced Endoscopists at various centers in the U.S, and outside U.S., use Choledochoscopy with SpyGlass to assist in the confirmation of diagnosis in patients having Billiary lesions. However, there is little data and thus neglibible evidence regarding the agreement of SPY interpretation within doctors. However, advanced endoscopists have only recently started to employ the SpyGlassTM Direct Visualization System for single operator choledochoscopy. Hence we lack enough data to accurately evaluate the sensitivity, specificity, accuracy, technical feasibility, safety and cost effectiveness of such imaging devices. Evaluation of these factors would help us compare them to conventional diagnostic options; and consequently help us identify appropriate imaging techniques for biliary and pancreatic disorders and improve clinical management of patients.

The purpose of this registry is to record information and evaluate the impact of SpyGlassTM Direct Visualization System for choledochoscopy on the management of pancreatico-biliary disorders. The registry will evaluate diagnostic performance and overall clinical management impacted by SpyGlass.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has undergone SpyGlass Choledochoscopy procedures for diagnosis and/or treatment of a pancreatico-biliary disorder
* Above 18 years of age

Exclusion Criteria:

* Any patient who has not undergone choledochoscopy for pancreatico-biliary disorders
* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who has undergone SpyGlass Choledochoscopy procedures for diagnosis and/or treatment of a pancreatico-biliary disorder
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-10; Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Management | 1 year
  Documentation of accuracy, sensitivity, specificity, positive predictive value, negative predictive value based on final diagnosis variable (followup at a year for confirmed diagnosis if tissue results are negative or indeterminate).

SECONDARY OUTCOMES:
Safety Profile | 30 days post procedure
  Documentation of Safety: Number of Participants with Adverse Events; Type, frequency and intensity of adverse events.

OTHER OUTCOMES:
Efficacy profile | 1 year
  Documentation of technical success and clinical success rates. Technical success is defined as successful choledochoscopy done or not based on access and visual recording.
  Clinical success is defined as determination of diagnosis based on choledochoscopy imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No IPD sharing

REFERENCES:
- [Derived] Kahaleh M, Gaidhane M, Shahid HM, Tyberg A, Sarkar A, Ardengh JC, Kedia P, Andalib I, Gress F, Sethi A, Gan SI, Suresh S, Makar M, Bareket R, Slivka A, Widmer JL, Jamidar PA, Alkhiari R, Oleas R, Kim D, Robles-Medranda CA, Raijman I. Digital single-operator cholangioscopy interobserver study using a new classification: the Mendoza Classification (with video). Gastrointest Endosc. 2022 Feb;95(2):319-326. doi: 10.1016/j.gie.2021.08.015. Epub 2021 Aug 31. PMID 34478737
- [Derived] Kahaleh M, Raijman I, Gaidhane M, Tyberg A, Sethi A, Slivka A, Adler DG, Sejpal D, Shahid H, Sarkar A, Martins F, Boumitri C, Burton S, Bertani H, Tarnasky P, Gress F, Gan I, Ardengh JC, Kedia P, Arnelo U, Jamidar P, Shah RJ, Robles-Medranda C. Digital Cholangioscopic Interpretation: When North Meets the South. Dig Dis Sci. 2022 Apr;67(4):1345-1351. doi: 10.1007/s10620-021-06961-z. Epub 2021 Mar 30. PMID 33783691